CLINICAL TRIAL: NCT05198102
Title: To Evaluate the Immunogenicity and Safety of Booster Immunization 12 Months After the Completion of Basic Immunization of Recombinant Novel Coronavirus Vaccine (CHO Cell) in People 18 Years Old and Above
Brief Title: ZF2001 Booster Immunization Clinical Trials of 12 Months After the Completion of Basic Immunization
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2021-NCV-JQ02
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-01

CONDITIONS: Prevention of COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational vaccine group (Experimental): Recombinant novel coronavirus vaccine (CHO cells) injection, Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person dose.
  Interventions: Biological: Recombinant novel coronavirus vaccine (CHO cells)

INTERVENTIONS:
Biological: Recombinant novel coronavirus vaccine (CHO cells) — At 12 months after the basic immunization (window period ± 3 months), 1 dose of recombinant novel coronavirus vaccine (CHO cells) is vaccinated.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the recombinant novel coronavirus vaccine (CHO cells) after the booster immunization. It is planned to screen 300 subjects of 18 years old and above who have completed the basic immunization of recombinant novel coronavirus vaccine (CHO cells), to evaluate the immunogenicity and safety of the booster immunization of 12 months (window period ± 3 months) after the basic immunization. Investigate the geometric mean titer (GMT), GMI and 4 times growth rate of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody 14 days, 30 days, and 6 months after booster vaccination; the incidence of all AEs within 1 month after the booster vaccination, the incidence of all serious adverse events (SAE) within 6 months after the booster vaccination.

DETAILED DESCRIPTION:
This study adopts an open experimental design. It is planned to screen 300 subjects of 18 years old and above who have completed the basic immunization of recombinant novel coronavirus vaccine (CHO cells), to evaluate the immunogenicity and safety of the booster immunization of 12 months (window period ± 3 months) after the basic immunization.

Immunogenicity observation: the geometric mean titer (GMT), GMI and 4 times growth rate of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody 14 days, 30 days, and 6 months after booster vaccination.

Safety observation:

All adverse events (AE) were collected within 30 minutes after the booster immunization, all AEs (including both solicited and unsolicited AEs) 0-7 days after the booster immunization, and all AEs (unsolicited AEs) 8-30 days after the booster immunization.

Solicited AE (the following events occurring within 7 days of vaccination) :

Adverse events at the inoculation site (local) : pain, pruritus, redness, swelling, rash, induration; Non-inoculated site (systemic) adverse events: fever, headache, fatigue, diarrhea, nausea, vomiting, muscle pain (non-inoculated site), acute allergic reactions, cough.

All SAEs were collected within 6 months after the booster immunization.

ELIGIBILITY:
Inclusion Criteria:

* Participated in "A Phase III Randomized, Double-blind, Placebo-controlled Clinical Trial in 18 Years of Age and Above to Determine the Safety and Efficacy of ZF2001, a Recombinant Novel Coronavirus Vaccine (CHO cell) for Prevention of COVID-19. Protocol no.: LKM-2020-NCV-GJ01)" and has completed basic immunization with recombinant novel coronavirus vaccine (CHO cells) since 12 months (window period ± 3 months);
* The subjects voluntarily participate in the study, sign an informed consent form, and can provide valid identification, understand and comply with the requirements of the trial protocol;
* Female subjects of childbearing age agree to take effective contraceptive measures from the start of the study to 1 month after vaccination.

Exclusion Criteria:

* A confirmed case of new coronavirus infection or asymptomatic infection or a history of positive new coronavirus nucleic acid test;
* Patients with uncontrolled lymphoproliferative diseases, unresolved aplastic anemia, active primary immune thrombocytopenia (ITP), uncontrolled coagulopathy, etc;
* Patients with malignant tumors before and after surgery, patients undergoing chemotherapy, radiotherapy, immunotherapy, etc.; patients with organ transplant status;
* People with uncontrolled epilepsy and other serious neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.);
* Suffering from acute diseases, or acute attacks of chronic diseases, or uncontrolled severe chronic diseases, such as hypertension that cannot be controlled by drugs (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg);
* Previous history of severe allergies to any vaccine, or history of severe allergies to any component of the test vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, dyspnea, vascular nerve Sexual edema, etc.;
* Women who are breastfeeding or pregnant;
* In addition to completing the recombinant new coronavirus vaccine (CHO cell) within the past 15 months, has participated in or is participating in other COVID-19 related clinical trials;
* Researchers believe that any disease or condition in the subject may put the subject at an unacceptable risk; the subject cannot meet the requirements of the protocol; the situation that interferes with the assessment of the vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Immunogenicity endpoint | 14 days after booster vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody
Immunogenicity endpoint | 30 days after booster vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody
Immunogenicity endpoint | 6 months after booster vaccination
  Geometric mean titer (GMT) of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody

SECONDARY OUTCOMES:
Immunogenicity endpoint | 14 days, 30 days, and 6 months after booster vaccination
  GMI and 4 times growth rate of SARS-CoV-2 neutralizing antibody and RBD protein binding antibody
Safety endpoint | Within 1 month after booster vaccination
  Incidence of all AEs
Safety endpoint | Within 6 months after booster vaccination
  Incidence of all SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Bachelor, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No